CLINICAL TRIAL: NCT01397123
Title: The Impact of an Intervention Taught by Trained Teachers on Childhood BMI z Score
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minho (Other)
Collaborators: Universidade do Porto (Other)
Responsible Party: Rafaela Rosário, University of Minho
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Prevention
Other Study IDs: 1845; 7613/2008 (Other: Portuguese Data Protection Authority)
Record Dates: First submitted 2011-06-28; First posted 2011-07-19 (Estimated); Last update posted 2011-07-19 (Estimated); Status verified 2011-07

CONDITIONS: Evidence of an Intervention on Childhood BMI z Score
Keywords: BMI z-score; children; overweight; school-based intervention; trained teachers; fruit; vegetables; Low nutrition energy dense foods
MeSH Terms: conditions — Overweight

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Lifestyle counseling (Experimental)
  Interventions: Other: Training teachers on healthier lifestyles

INTERVENTIONS:
Other: Training teachers on healthier lifestyles — During 2007/2008 seven out of eighty public elementary public schools from Guimarães (Portugal) were invited to participate in this study. The number of schools involved was according to constraints of personnel for the assessment and intervention. Schools were the unit of randomization and three were assigned into intervention, and four into control group. Data was collected prior to intervention and immediately after, during the year 2009 (post-intervention). Prior to participation on data collection, parents provided informed consent, and children provided oral assent.

SUMMARY:
The purpose of this study is to assess the effects of a six months nutrition intervention, delivered and taught by classroom teachers with in-service nutrition training, on the prevention of overweight and obesity among children in grades 1 to 4.

In this randomized controlled trial, 464 children from seven elementary schools were allocated to a six months nutrition educational intervention by their own teachers or to standard care. Intervened teachers had 12 sessions of three hours each with the researchers throughout six months, according to the following topics: nutrition and healthy eating (sessions 1 to 4); the importance of drinking water (session 5); strategies to encourage fruits and vegetables consumption and to decrease high energy-density foods intake (sessions 6 to 8); strategies to increase physical activity (sessions 9 and 10); and healthy cooking activities (sessions 11 and 12). After each session, teachers were encouraged to develop activities in class that focused on the learned topics. Sociodemographic, anthropometric, dietary, and physical activity assessments were performed at baseline and the end of intervention.

We expect that fewer intervened children become overweight and the consumption of fruit and vegetables will be higher. In addition, we expect a less consumption of low-nutrition high dense foods.

We also expect to provide further support to decrease overweight epidemic, involving classroom teachers in a training intervention and making them dedicated interventionists.

DETAILED DESCRIPTION:
The prevalence of obesity continues to increase (Ogden et al., 2006) and is growing concerns in Portugal and in the world. As successful treatments have been elusive, the prevention should be considered a high priority. So, present efforts are being dedicated to develop and implement overweight and obesity prevention interventions (Gortmaker, et al, 1999; James, Tomas & Kerr, 2004), in the hope that multilevel approach, if occur early in childhood, may improve eating habits and physical activity and therefore, contribute to prevent or reverse this epidemic state.

In each school, previously trained persons performed anthropometric evaluation, using standardized procedures (WHO Expert Commitee 1995). Anthropometric measurements were performed in children with light indoor clothing and barefooted. Weight was measured in an electronic scale, with an error of ±100g (Seca, Model 703, Germany), and height was measured using a stadiometer, with the head in the Frankfort plane. BMI was computed as mass, Kg/height, m2. The prevalence of underweight, normal weight, overweight and obesity was calculated according to the International Obesity Task Force (IOTF) criteria, making a correspondence between the traditional adult cut-off and specific values for children according to gender and age (Cole et al. 2000). A z-score (the number of standard deviations (SD) from the reference population) was calculated for each child using the LMS method and the calculation was determined using the LMS growth add-in for excel (Pan and Cole 2009).

Dietary intake was gathered by 24h dietary recalls obtained by nutritionists and/or trained interviewers. We assessed a single recall before and another after the intervention. The respondents had no prior notification of when the recalls would occur. Training of interviewers included practice using photos and food models to quantify portion sizes, experience in probing information from children without suggesting responses as well as the type of food consumed in detail of fat content, brand name, constituents of mixed dishes and so on. The 24h dietary recall is the most commonly used dietary assessment method because it is easy to administer, can be performed in large-scale studies (Kranz and Sie-Riz 2002, Gomez-Martínez et al. 2009), and can be used to assess adequacy of energy and macronutrient intakes. During the 24h dietary recall, each child was asked to recall all food and beverages consumed during the past 24h. Daily routines were used as prompts (waking up, going to bed, time between classes, and before or after school) to enhance recall. Portion sizes of foods and beverages consumed were also estimated using food models, photos and other props (cups, glasses, food wrappers or containers) as an aid in determining serving sizes. Energy and nutritional intake were estimated using an adapted Portuguese version of the nutritional analysis software Food Processor Plus (ESHA Research Inc., Salem, OR, USA). The 24-hour dietary recall interviews captured the time and name of each eating occasion, the foods and beverages reported at each eating occasion, and the source from which item was obtained.

In order to assess the level of physical activity of children, parents were asked five questions with four answer choices (4-point scale) ranging from 0 (very seldom) to 4 (very often): a) Outside the school does your child take part in organized sport? b) Outside school does your child take part in non-organized sport? c) Outside school, how many times a week does your child take part in sport or physical activity for at least 20 minutes? d) Outside school hours, how many hours a week does your child usually take part in physical activity so much that he gets out of breath or sweat? e) Does your child take part in competitive sport? (Mota and Esculcas 2002). The total sum of the points was computed reaching a maximum of 20 points. To express the activity levels, a Physical Activity Index was obtained, which divided the sample into four activity classes: sedentary group (0-5); low activity group (6-10); moderately active group (11-15); and vigorously active group (16-20), on the basis of their reported physical activity (Mota and Esculcas 2002).

Social, demographic and family characteristics were assessed by questionnaire. The survey sent to parents contained questions about gender and age of children, education of the parents (recorded in five categories: 0, 1-4, 5-9, 10-12, and more than 12 years of formal education). This information was further grouped for analysis into three categories: up to 9 years, 10-12 years, and more than 12 years of education.

The research team proposed, in January 2008, the accreditation of the sessions that were developed with the teachers to the Minister of Education, Scientific-Pedagogic Council for In-service Training (Conselho Científico Pedagógico da Formação Contínua, Ministério da Educação). This proposal was approved in September 2008 in the form of "training workshop" with 72 hours duration, distributed by active learning strategies (36 hours) and work contact with the children (36 hours). Teachers of the intervention group had 12 sessions of three hours each with the researchers throughout six months, which included the following topics: nutrition and healthy eating for the children and the families (sessions 1 to 4); the importance of the water (session 5); strategies to encourage fruits and vegetables consumption and to decrease high energy density foods intake (sessions 6 to 8); to increase physical activity and to reduce screen time exposure (sessions 9 and 10); and healthy cooking (sessions 11 and 12). After each session, teachers resend the learned contents to develop creative and engaging classroom activities about the addressed topic. All the questions that arose during the implementation of classroom activities were addressed and resolved shortly with the researchers. Teachers were allowed to develop and refine the activities and learning strategies that were proposed by researchers. At the end of this period, the teachers delivered a critical report of activities focused on the work contact with children.

The data analysis was performed using SPSS ®, Version 18.0 (SPSS Inc; Chicago, IL).

ELIGIBILITY:
Inclusion Criteria:

* Children from the schools involved in the study with informed consent provided by parents.

Exclusion Criteria:

* Age more than 12

Ages: 5 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 464 (Actual)
Dates: Start 2007-09; Primary Completion 2008-06 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
BMI z score | the first 3 months after the intervention

SECONDARY OUTCOMES:
dietary intake | within the first 3 months after the intervention

CONTACTS AND LOCATIONS:
Overall Officials: Pedro Moreira, PhD, Study Director — Universidade do Porto; Beatriz Pereira, PhD, Study Director — University of Minho; Rafaela V Rosario, Principal Investigator — University of Minho
Locations (1):
- Santos Simões group of schools, Guimarães, Braga District, Portugal

REFERENCES:
- [Background] Cole TJ, Bellizzi MC, Flegal KM, Dietz WH. Establishing a standard definition for child overweight and obesity worldwide: international survey. BMJ. 2000 May 6;320(7244):1240-3. doi: 10.1136/bmj.320.7244.1240. PMID 10797032
- [Background] Kranz S, Siega-Riz AM. Sociodemographic determinants of added sugar intake in preschoolers 2 to 5 years old. J Pediatr. 2002 Jun;140(6):667-72. doi: 10.1067/mpd.2002.124307. PMID 12072868
- [Background] Ogden CL, Carroll MD, Curtin LR, McDowell MA, Tabak CJ, Flegal KM. Prevalence of overweight and obesity in the United States, 1999-2004. JAMA. 2006 Apr 5;295(13):1549-55. doi: 10.1001/jama.295.13.1549. PMID 16595758
- [Background] Goldberg GR, Black AE, Jebb SA, Cole TJ, Murgatroyd PR, Coward WA, Prentice AM. Critical evaluation of energy intake data using fundamental principles of energy physiology: 1. Derivation of cut-off limits to identify under-recording. Eur J Clin Nutr. 1991 Dec;45(12):569-81. PMID 1810719
- [Background] Gomez-Martinez S, Martin A, Romeo J, Castillo M, Mesena M, Baraza JC, Jimenez-Pavon D, Redondo C, Zamora S, Marcos A. Is soft drink consumption associated with body composition? A cross-sectional study in Spanish adolescents. Nutr Hosp. 2009 Jan-Feb;24(1):97-102. PMID 19266121
- [Background] Mota J, Esculcas C. Leisure-time physical activity behavior: structured and unstructured choices according to sex, age, and level of physical activity. Int J Behav Med. 2002;9(2):111-21. doi: 10.1207/s15327558ijbm0902_03. PMID 12174530
- [Background] Schofield WN. Predicting basal metabolic rate, new standards and review of previous work. Hum Nutr Clin Nutr. 1985;39 Suppl 1:5-41. PMID 4044297
- [Derived] Rosario R, Araujo A, Padrao P, Lopes O, Moreira A, Pereira B, Moreira P. Health Promotion Intervention to Improve Diet Quality in Children. Health Promot Pract. 2017 Mar;18(2):253-262. doi: 10.1177/1524839916634096. Epub 2016 Jul 9. PMID 27095035